CLINICAL TRIAL: NCT06145256
Title: Radiological Evaluation of Hypoxic Ischemic Encephalopathy in Neonatal Intensive Care Unit Of Assuit University Children's Hospital
Brief Title: Radiological Evaluation of Hypoxic Ischemic Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Azab Abdelatty, Principal Investigator at Assuit University pediatric department, Assiut University
Other Study IDs: Radiological Evaluation of HIE
Record Dates: First submitted 2023-10-18; First posted 2023-11-24 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Hypoxic Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI brain, MSCT brain, Transcranial Ultrasound — MRI, MSCT and transcranial Ultrasound are an important diagnostic modalities in the assessment of severity and outcome of HIE

SUMMARY:
To compare between Transcranial Ultrasound , MRI and CT in patients with Hypoxic Ischemic Encephalopathyas regards diagnostic accuracy and prognostic value .

DETAILED DESCRIPTION:
* Hypoxic Ischemic Encephalopathy (HIE) is an injury to the brain, occurring in the neonatal period (under 28 days old) in which there is deprivation of oxygen supply to brain. It is a common cause of neonate mortality and developmental psychomotor disorders in the pediatric population worldwide.This is one of the major causes of cerebral palsy."
* Hypoxic ischemic encephalopathy (HIE) is one of the most serious birth complications affecting full term infants. It occurs in 1.5 to 2.5 per 1000 live births in developed countries and 2.3-26.5 per 1000 live births in developing countries . The incidence of HIE has not declined even with advances in obstetric care (i.e. fetal monitoring) aimed at preventing the hypoxicischemic event; thus much of the current neonatal research about HIE focuses on minimizing the extent of subsequent brain injury.
* HIE is a disorder in which clinical manifestations indicate brain dysfunction.While the exact cause is not always identified, antecedents include cord prolapse, uterine rupture, abruptio placenta, placenta previa, maternal hypotension, breech presentation, or shoulder dystonia. The manifestations of perinatal HIE in early postnatal life include abnormal fetal heart rate tracings, poor umbilical cord gases (pH < 0.7 or base deficit ≥ 12 mmol/L),low Apgar scores, presence of meconium stained fluid,or the need for respiratory support within the first several minutes of postnatal life.
* The infant usually develops seizure within first 24 h of life. Children with periventricular leukomalacia (PVL) may develop spastic CP in the form of diplegia, quadriplegia, or hemiplegia.Involvement of subcortical white matter produces severe mental retardation and impaired vision.Basal ganglia (BG) and thalamic involvement result in extrapyramidal symptoms. Multicystic encephalopathy is associated with quadriplegia, bulbar and choreoathetoid symptoms, microcephaly and mental retardation. Abnormal electroencephalographic (EEG) findings may predict adverse clinical outcome such as long-term neurologic sequelae or impending death.
* Multiple neuroimaging techniques are available to visualize brain injury in the neonatal period. Cranial ultrasonography is a helpful noninvasive tool to detect antenatal onset of injury and abnormalities that may mimic HIE. Abnormalities related to HIE can be recognized with ultrasonography as well, but it will take 48-72 h to see these changes develop in the white matter or deep gray nuclei . Magnetic resonance imaging (MRI) which includes diffusion-weighted imaging (DWI) is the preferred imaging modality during the first week after birth to determine the extent of brain injury and predict neurodevelopmental outcome in infants with symptoms of HIE, without its prognostic utility being altered by therapeutic hypothermia .
* CT image could be used as important diagnostic indication in the assessment of HIE neonate CT could identify subarachnoid hemorrhage. It is valuable in clinical application

ELIGIBILITY:
Inclusion Criteria:

* all term and preterm newborns who suffered perinatal asphyxia and all neonatal with clinical manifestations suggestive of hypoxic ischemic encephalopathy :

  1. disturbed level of consciousness
  2. low apgar score 3_ low pH in blood gases within the first hours of delivery 4_ neonatal seizures within first 48 h of delivery

Exclusion Criteria:

* Those newborns with :

  1. CNS infections
  2. sepsis
  3. respiratory distress
  4. metabolic disorders
  5. major congenital malformations Were excluded from the study

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * study population comprised of all term and preterm newborns who suffered perinatal asphyxia and all neonatal with clinical manifestations suggestive of hypoxic ischemic encephalopathy :
    1. disturbed level of consciousness
    2. low apgar score 3_ low pH in blood gases within the first hours of delivery 4_ neonatal seizures within first 48 h of delivery and excluded Those newborns with :
    <!-- -->
    1. CNS infections
    2. sepsis
    3. respiratory distress
    4. metabolic disorders
    5. major congenital malformations From the study
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
To determine how many children born with clinical suspicion of HIE actually have radiological findings corresponding to the clinical picture | one year
  To determine how many children born with clinical suspicion of HIE ( low apgar score , low pH in blood gases within first hours of delivery, disturbed level of consciousness and neonatal seizures ) actually have radiological findings corresponding with the clinical picture

REFERENCES:
- See also: Related Info — http://www.who.int/westernpacific/health-topics/newborn-health